CLINICAL TRIAL: NCT03072901
Title: Registry Observing EndoBarrier® Treatment Outcomes in Subjects With Type 2 Diabetes and/or Obesity
Status: Terminated | Type: Observational
Why Stopped: GID terminated the Registry due to evolving registry requirements
Sponsor: Morphic Medical Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-3
Record Dates: First submitted 2017-01-19; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- EndoBarrier Gastrointestinal Liner: 244 subjects; The registry will be open to subjects who meet the EndoBarrier's Indications for Use and none of the Contraindications in the device's Instructions For Use document. Subjects who successfully receive the device implant at a participating registry center will be included in the registry.
  Interventions: Device: EndoBarrier Gastrointestinal Liner

INTERVENTIONS:
Device: EndoBarrier Gastrointestinal Liner — The EndoBarrier Gastrointestinal Liner (EndoBarrier) is a nonsurgical metabolic intervention for the treatment of Type 2 diabetes and obesity. By bypassing the duodenum and proximal jejunum, the device may alter signaling pathways that control metabolic processes.1, 2 The effect on patient's glucose levels is immediate as evidenced by meal tolerance testing.3 Since the device also promotes reduced appetite resulting in weight loss, the effect is maintained as the patient loses weight over the implant period. Most patients achieve normal HbA1c and fasting plasma glucose (FPG) levels rapidly within 3-6 months.

SUMMARY:
The purpose of the registry was to observe the safety and effectiveness outcomes for subjects treated with the EndoBarrier in the post market setting where the product had Conformité Européene (CE mark) regulatory approval and in accordance to the approved Indication For Use.

DETAILED DESCRIPTION:
This was a worldwide observational registry of the use of the EndoBarrier for inclusion of subjects treated with the EndoBarrier in centers in Australia, Chile, and the Netherlands. The registry was open to all subjects at participating centers that received the EndoBarrier.

ELIGIBILITY:
Inclusion Criteria:

* As per IFU, the EndoBarrier GI liner System is used for the treatment of obese type 2 diabetes with BMI greater than or equal to 30 kg/m2, or obese patients with BMI greater than or equal to 30 kg/m2 with less than or equal to 1 co-morbidities, or obese patients with BMI greater than 35 kg/m2. The GI liner is indicated for a maximum implant duration of 12 months.

Exclusion Criteria:

As per Instructions For Use (IFU)

* Women who are pregnant
* Requirement for prescription anticoagulation therapy
* History of inflammatory bowel disease or condition of the gastrointestinal tract, such as peptic ulcer disease (PUD), ulcers, or Crohn's disease
* Pancreatitis, Uncontrolled gastroesophageal reflux disease (GERD), Known infection at the time of implant
* Symptomatic coronary artery disease or pulmonary dysfunction
* History of coagulopathy
* Bleeding diathesis, upper GI bleeding conditions such as esophageal or gastric varices, or congenital or acquired intestinal telangiectasia
* Congenital or acquired anomalies of the GI tract such as atresias or stenosis
* Previous GI surgery that could affect the ability to place the EndoBarrier Gastrointestinal Liner or its function
* Iron deficiency and/or iron deficiency anemia
* Active symptoms of kidney stones or known presence of gallstones
* Inability to discontinue use of non-steroidal anti-inflammatory drugs during the implant period
* Family or patient history of known diagnosis or pre-existing condition of systemic lupus erythematosus, scleroderma, or other autoimmune connective tissue disorder
* H. pylori positive status (Patients may receive the EndoBarrier Gastrointestinal Liner if they had a prior history and were successfully treated)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry was open to subjects who met the EndoBarrier's Indications for Use, inclusion/exclusion criteria and contraindications in the device's Instructions For Use at the time the Registry was initiated.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2010-12; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 24 months
Evaluation of Effectiveness of the EndoBarrier GI Liner upon glycemic control | Change from Baseline measured up to 24 months
  Change in %HbA1c from Baseline
Evaluation of Effectiveness of the EndoBarrier GI Liner upon weight loss | Change from Baseline measured up to 24 months
  Change from Baseline of weight (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Gersin, MD, Study Director — GI Dynamics, Medical Director

IPD SHARING:
Plan to Share IPD: No